CLINICAL TRIAL: NCT04162366
Title: Multi-center, Blinded, Randomized Study With Aprocitentan in Subjects With Uncontrolled Blood Pressure and Chronic Kidney Disease Stage 3 or 4.
Brief Title: A Research Study to Show Aprocitentan is Efficacious and Safe to Treat Patients With Uncontrolled Blood Pressure and Chronic Kidney Disease.
Acronym: INSPIRE-CKD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: A business decision was made to not initiate this study
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-080A305; 2018-003819-22 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Hypertension; Renal Insufficiency, Chronic
Keywords: Chronic kidney disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — aprocitentan

STUDY DESIGN:
Intervention Model Description: All participants will get the active drug, aprocitentan 25 mg, for at least 8 weeks. All participants will receive placebo for 2 weeks. During a certain period of the study, participants will receive aprocitentan 25 mg or placebo for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aprocitentan 25 mg (Experimental)
  Interventions: Drug: Aprocitentan 25 mg
- Placebo (Experimental)
  Interventions: Drug: Placebo
- Aprocitentan 25 mg or Placebo (Experimental)
  Interventions: Drug: Aprocitentan 25 mg; Drug: Placebo

INTERVENTIONS:
Drug: Aprocitentan 25 mg — Tablet, oral use once daily
  Other Names: ACT-132577
  Arms: Aprocitentan 25 mg; Aprocitentan 25 mg or Placebo
Drug: Placebo — Matching placebo tablet, oral use once daily
  Arms: Aprocitentan 25 mg or Placebo; Placebo

SUMMARY:
The purpose of this research study is to show the blood pressure lowering effect of aprocitentan, a new drug, when added to the background antihypertensive therapy in patients with uncontrolled blood pressure and chronic kidney disease (CKD) stage 3 or 4. Participation in the research study will last up to 21 weeks (about 5 months).

ELIGIBILITY:
Inclusion Criteria:

* Prior treatment with at least 2 anti-hypertensive medications, at optimal or best tolerated dose, of different pharmacological classes, including a diuretic,
* Participants with uncontrolled blood pressure (mean sitting systolic blood pressure of 140 mmHg or greater) and chronic kidney disease stage 3 or 4 (estimated Glomerular Filtration Rate of at least 15 and below 60 mL/min/1.73m2 using the Chronic Kidney Disease-Epidemiology equation),
* Women of childbearing potential are eligible only if the following applies:

  * Negative pregnancy test at the screening visit and at baseline (i.e., end of run-in period).
  * Agree to undertake pregnancy tests during the study and up to 30 days after randomized study treatment discontinuation.
  * Agree to use highly-effective methods of contraception up to at least 30 days after study treatment discontinuation.

Exclusion Criteria:

* Mean sitting systolic blood pressure above 170 mmHg measured by "automated office blood pressure measurement" (AOBPM),
* Mean sitting diastolic blood pressure above 105 mmHg measured by AOBPM,
* Change in renal function requiring hospitalization, documented eGFR decline of greater than 20% in the 3 months prior to the screening visit, dialysis in the 3 months before the screening visit,
* Planned dialysis or kidney transplant during the course of this study,
* Nephrotic syndrome defined as urine albumin-to-creatinine ratio above 3000 mg/g,
* Known and documented chronic heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 of double-blind treatment in mean trough sitting systolic blood pressure measured by automated office blood pressure measurement. | From baseline to Week 4 after treatment initiation

SECONDARY OUTCOMES:
Change from baseline to Week 4 of double-blind treatment in mean trough sitting diastolic blood pressure measured by automated office blood pressure measurement. | From baseline to Week 4 after treatment initiation
Ratio to baseline of urine albumin-to-creatinine ratio (UACR) at Week 4 | From baseline to Week 4 after treatment initiation
  Evaluated in the subgroup of participants with a UACR greater than 30 mg/g at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.

IPD SHARING:
Plan to Share IPD: No